CLINICAL TRIAL: NCT06949696
Title: Effects of Dual-Task Training and Cognitive Rehabilitation on Gait, Balance, Fatigue and Cognitive Performance in Individuals With Multiple Sclerosis
Brief Title: Effect of Dual-Task Training and Cognitive Rehabilitation in Individuals With Multiple Sclerosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Aysun Katmerlikaya, Research Assistant, Toros University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU-FTR-AK-01
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; balance; gait; dual task; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Comparison of 3 different physiotherapy groups(dual task training group, cognitive rehabilitation group, conventional physical therapy group)
Who Masked: Outcomes Assessor
Masking Description: A randomized, single-blind, controlled trial comparing a dual-task training group, a cognitive rehabilitation group, and a conventional physical therapy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual Task Training Group (Experimental): The dual task training group will receive training 2 days a week for 6 weeks. Patients will receive dual task training. They will also receive 30 minutes of individual physiotherapy exercises. 2 days a week. The effects of dual task training and cognitive rehabilitation on gait, balance, fatigue and cognitive performance will be compared.
  Interventions: Other: Dual Task Training
- Cognitive Rehabilitation Group (Experimental): The cognitive rehabilitation group will receive training 2 days a week for 6 weeks. Patients will receive cognitive rehabilitation group. They will also receive 30 minutes of individual physiotherapy exercises 2 days a week.
  Interventions: Other: Cognitive Rehabilitation
- Conventionel Physiotherapy Group (Active Comparator): The conventionel physiotherapy group will receive training 2 days a week for 6 weeks.This group will only receive individual physiotherapy 2 days a week.
  Interventions: Other: Conventionel Physiotherapy

INTERVENTIONS:
Other: Dual Task Training — In dual task training, patients will be given cognitive exercises such as counting backwards from 100 by 3, counting the names of cities, girls and boys while walking.
  Arms: Dual Task Training Group
Other: Cognitive Rehabilitation — In cognitive rehabilitation, patients will be given paper-and-pencil activities and exercises to find the difference between two pictures.
  Arms: Cognitive Rehabilitation Group
Other: Conventionel Physiotherapy — In conventionel physiotherapy, patients will be given posture exercises for balance and strengthening.
  Arms: Conventionel Physiotherapy Group

SUMMARY:
The purpose of this study is to examine the effects of dual-task training and cognitive rehabilitation on gait, balance, fatigue and cognitive performance in individuals with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a complex disease characterized by chronic, inflammatory, demyelinating and neurodegenerative processes of the central nervous system (CNS) with heterogeneous clinical symptoms. Balance, gait and cognitive impairment are among the biggest problems in individuals with MS and significantly affect their daily lives.

Dual Task (DT); is the process of performing two tasks that can be performed independently and have different purposes simultaneously. Walking with dual tasks has recently been shown to resemble typical walking performance in daily life, thus providing clinicians with a realistic walking performance measurement in daily life. Although the effects of dual task performance in various neurological diseases have been partially described in the literature, the comparison of dual task training and cognitive rehabilitation on walking, balance, fatigue and cognitive performance has not been made and due to this deficiency in the literature, our study was planned and has originality. The aim of our study is to investigate the effects of dual task training and cognitive rehabilitation on walking, balance, fatigue and cognitive performance in individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis by a neurologist
* Can walk independently
* Expanded Disability Status Scale (EDSS) score below 5
* Has not had an attack in the last 3 months, has been medically stable for 6 months
* Has not received a regular physiotherapy program in the last 6 months volunteer

Exclusion Criteria:

* Scoring 26 or below on the Montreal Cognitive Assessment Scale (MoCA)
* Having systemic, orthopedic and neurological problems that may affect walking and balance in the assessments
* Having additional psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index (DGI) | a year
  DGI is a test that measures the capacity to adapt to changes in walking.It evaluates a total of 8 parameters over 24 points. Values of 19 points and below define the presence of a fall risk.

SECONDARY OUTCOMES:
Timed 25 Food Walk Test (T25FWT) | a year
  Timed 25 Food Walk Test is a test that evaluates walking speed. In the test, the patient is asked to walk 25 steps as quickly and safely as possible and the time is recorded in seconds with the average of 2 trials.
The 12-item MS Walking Scale (12-MSWS) | a year
  The 12-item MS Walking Scale (12-MSWS) that evaluates walking ability over the last 2 weeks, scaled from 0 to 100.
BICAMS (Brief International Cognitive Assessment for MS) | a year
  BICAMS (Brief International Cognitive Assessment for MS) is an international initiative to recommend and support a cognitive assessment that is brief, practical and universal.
Trial Making Test (TMT) | a year
  Trial Making Test (TMT)is used to evaluate individuals' executive functions, visual-motor perception, visual scanning and attention speed, motor function, organization, and planning.
Modified Fatigue Impact Scale (MFIS) | a year
  It is a multidimensional self-report questionnaire consisting of 21 questions in total, which is frequently used in individuals with MS and evaluates subjective fatigue physically (9 items), cognitively (10 items) and psychosocially (2 items).

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Katmerlikaya, MSc, Principal Investigator — Toros University; Öznur Tunca, Prof.Dr., Study Director — Hacettepe University; Serhan Sevim, Prof.Dr., Study Chair — Mersin University; Yeliz Salcı, Assoc.Prof., Study Chair — Hacettepe University; Dilek Hande Esen, PhD, Study Chair — Toros University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozkul C, Guclu-Gunduz A, Eldemir K, Apaydin Y, Gulsen C, Yazici G, Soke F, Irkec C. Dual-Task Cost and Related Clinical Features in Patients With Multiple Sclerosis. Motor Control. 2021 Jan 12;25(2):211-233. doi: 10.1123/mc.2020-0035. PMID 33440347
- [Result] Abasiyanik Z, Kahraman T. Effect of dual-task training on cognitive functions in persons with multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2022 Jun;62:103801. doi: 10.1016/j.msard.2022.103801. Epub 2022 Apr 10. PMID 35430546
- See also: Effect of dual-task training on cognitive functions in persons with multiple sclerosis: A systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/35430546/
- See also: Dual-Task Cost and Related Clinical Features in Patients With Multiple Sclerosis — https://pubmed.ncbi.nlm.nih.gov/33440347/